CLINICAL TRIAL: NCT04538599
Title: RD13-01 for Patients With r/r CD7+ T/NK Cell Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, PhD, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD13-01-02
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-09

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-01 cell infusion (Experimental)
  Interventions: Drug: RD13-01 cell infusion

INTERVENTIONS:
Drug: RD13-01 cell infusion — Universal CAR-T cells targeting CD7

SUMMARY:
This study is designed to explore the safety of RD13-01 for patients with CD7+ relapsed and/or refractory T/NK-cell hematologic malignancies. And to evaluate the efficacy and pharmacokinetics of RD13-01 in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3 to 70 years.
2. Diagnosis of r/r T-ALL/NK-ALL, T-LBL, or T-NHL (including PTCL-NOS, AITL, ALCL, Extranodal NK/T cell lymphoma).
3. ECOG: 0-2.
4. Life expectancy greater than 12 weeks.
5. Cardiac left ventricle ejection fraction ≥50%.
6. Informed consent explained to, understood by and signed by the patient/guardian. Patient/guardian is given a copy of informed consent.

Exclusion Criteria:

1. Pregnant or lactating.
2. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Viral (HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA positive; syphilis positive.
3. Patients with graft-versus-host disease (GVHD) or who need to use immunosuppressive drugs.
4. Participated in other clinical studies within 2 weeks prior to screening.
5. History of alcoholism, drug abuse or mental illness.
6. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 4 weeks after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Hu Y, Zhang M, Yang T, Mo Z, Wei G, Jing R, Zhao H, Chen R, Zu C, Gu T, Xiao P, Hong R, Feng J, Fu S, Kong D, Xu H, Cui J, Huang S, Liang B, Yuan X, Cui Q, Guo H, Yu Y, Feng Y, Jin C, Ren J, Chang AH, Wang D, Huang H. Sequential CD7 CAR T-Cell Therapy and Allogeneic HSCT without GVHD Prophylaxis. N Engl J Med. 2024 Apr 25;390(16):1467-1480. doi: 10.1056/NEJMoa2313812. PMID 38657244
- [Derived] Hu Y, Zhou Y, Zhang M, Zhao H, Wei G, Ge W, Cui Q, Mu Q, Chen G, Han L, Guo T, Cui J, Jiang X, Zheng X, Yu S, Li X, Zhang X, Chen M, Li X, Gao M, Wang K, Zu C, Zhang H, He X, Wang Y, Wang D, Ren J, Huang H. Genetically modified CD7-targeting allogeneic CAR-T cell therapy with enhanced efficacy for relapsed/refractory CD7-positive hematological malignancies: a phase I clinical study. Cell Res. 2022 Nov;32(11):995-1007. doi: 10.1038/s41422-022-00721-y. Epub 2022 Sep 23. PMID 36151216